CLINICAL TRIAL: NCT00472524
Title: Cycloplegic Delivery Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2003H0072
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Healthy

INTERVENTIONS:
Procedure: Mydriasis/cycloplegia via different modes of administration

SUMMARY:
The goal of this study is to compare the effectiveness of the administration of sequential drops, a combination drop and a combination spray for producing mydriasis and cycloplegia.

ELIGIBILITY:
Inclusion Criteria:

* patients ages 8 to 30 with best corrected acuity of 20/30 or better in both eyes at distance and near will be recruited.

Exclusion Criteria:

* vision not correctable to 20/30 or better

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50

CONTACTS AND LOCATIONS:
Overall Officials: Marjean Kulp, OD, MS, Principal Investigator — Ohio State University